CLINICAL TRIAL: NCT01220258
Title: A Single-Center, Open-Label Study to Characterize Eyelid Margin Erythema, Markers of Clinical Inflammation and Levels of Inflammatory Mediators in the Lid Margins and Conjunctivae of Untreated Healthy Volunteers and Subjects Diagnosed With Posterior Blepharoconjunctivitis Following Dosing With Azithromycin Ophthalmic Solution, 1% for Four Weeks
Brief Title: A Four Week, Open-Label Study of Azithromycin Ophthalmic Solution, 1% (P08641)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08641; 041-118
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Posterior Blepharoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin ophthalmic solution, 1% (Experimental)
  Interventions: Drug: Azithromycin ophthalmic solution, 1%

INTERVENTIONS:
Drug: Azithromycin ophthalmic solution, 1% — 1 drop twice daily (BID) for the first 2 days and then 1 drop once daily (QD) for the remainder of treatment period (approximately 28 days total)

SUMMARY:
One objective of this study is to determine the levels of markers of inflammation on the eyelid margin of subjects with blepharoconjunctivitis and compare them with those of healthy volunteers. Another objective is to determine in subjects with blepharoconjunctivitis the effect of azithromycin ophthalmic solution, 1 % on markers of inflammation of lid margins and conjunctivae and on signs and symptoms of blepharoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of posterior blepharoconjunctivitis in both eyes

(except for healthy volunteers)

* Have a Best Corrected Visual Acuity (BCVA), using corrective lenses if necessary, in both eyes of at least +0.7 LogMAR
* If female, are non-pregnant or non-lactating

Exclusion Criteria:

* Have anterior blepharitis
* Have lid structural abnormalities
* Have had penetrating intraocular surgery in the past 90 days or require

penetrating intraocular surgery during the study

* Unable to withhold the use of contact lenses within 3 days prior to Visit 1

during the study

* Have been diagnosed with ongoing glaucoma
* Have a serious medical condition which could confound study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline of investigator-rated scores for eyelid margin erythema | Week 4

SECONDARY OUTCOMES:
Change from baseline of investigator-rated scores of blepharoconjunctivitis signs | Weeks 2, 4, 6, 8
Change from baseline of subject-rated scores of blepharoconjunctivitis symptoms | Weeks 2, 4, 6, 8

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, PhD, Study Chair — Medical Monitor
Locations (1):
- Baylor Eye Clinic, Alkek Eye Center of Baylor College of Medicine, Houston, Texas, United States